CLINICAL TRIAL: NCT00142935
Title: Opiate Replacement Therapy at Release From Incarceration
Brief Title: Effectiveness of Opiate Replacement Therapy Administered Prior to Release From a Correctional Facility - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIDA-18641-1; R01-DA018641-1; DPMC; R01DA018641 (NIH)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2009-05

CONDITIONS: HIV Prevention; Opioid-Related Disorders
Keywords: HIV Prevention; Opioid-Related Disorders; Medication Assisted Treatment; Methadone
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pre-Release Initiation MMT (Experimental): Participants assigned to this arm will undergo extensive assessment (physical, medical history, drug use and treatment history) prior to initiating treatment. MMT will begin 1-30 days prior to release from incarceration. MMT first dose will begin at 5 mg with 2 mg increase per day until release or therapeutic dose of 60-120 mg is achieved. Daily observation by dosing nurses and twice weekly symptom review by Research Assistant will occur. Additionally, participants assigned to Arm 1 will have all logistical arrangements made for entry into a community methadone clinic program within 24 hours of release from incarceration. The study will fully pay for MMT for 12 weeks and half the costs of treatment for the next 12 weeks.
  Interventions: Behavioral: Pre-release Initiation of MMT
- Post Release Initiation of MMT (Experimental): Participants assigned to this arm will have all logistical arrangements made for entry into a community methadone clinic program within 24-48 hours of release from incarceration. The study will fully pay for MMT for 12 weeks and half the costs of treatment for the next 12 weeks.
  Interventions: Behavioral: Post Release Initiation of MMT.
- Standard of Care Plus (Active Comparator): Participants assigned to this arem will not begin treatment prior to release from incarceration or have treatment paid for by the study. However, study staff will work with participants to identify ways to pay for treatment, including assisting with medicaid applications, etc. Further, the study will make the logistical arrangements for entering treatment if participant has a means to finance MMT.
  Interventions: Behavioral: Standard of Care Plus

INTERVENTIONS:
Behavioral: Pre-release Initiation of MMT — Participants assigned to arm 1 will undergo extensive assessment (physical, medical history, drug use and treatment history) prior to initiating treatment. MMT will begin 1-30 days prior to release from incarceration. MMT first dose will begin at 5 mg with 2 mg increase per day until release or therapeutic dose of 60-120 mg is achieved. Daily observation by dosing nurses and twice weekly symptom review by Research Assistant will occur. Additionally, participants assigned to Arm 1 will have all logistical arrangements made for entry into a community methadone clinic program within 24 hours of release from incarceration. The study will fully pay for MMT for 12 weeks and half the costs of treatment for the next 12 weeks.
  Arms: Pre-Release Initiation MMT
Behavioral: Post Release Initiation of MMT. — Participants assigned to Arm 2 will have all logistical arrangements made for entry into a community methadone clinic program within 24-48 hours of release from incarceration. The study will fully pay for MMT for 12 weeks and half the costs of treatment for the next 12 weeks.
  Arms: Post Release Initiation of MMT
Behavioral: Standard of Care Plus — Participants assigned to Arm 3 will not begin treatment prior to release from incarceration or have treatment paid for by the study. However, study staff will work with participants to identify ways to pay for treatment, including assisting with medicaid applications, etc. Further, the study will make the logistical arrangements for entering treatment if participant has a means to finance MMT.
  Arms: Standard of Care Plus

SUMMARY:
Much of the HIV/AIDS epidemic is driven by transmission from or to persons addicted to opiates. Many of these individuals pass through a correctional setting each year, creating an opportunity for linkage to substance abuse treatment. The purpose of this study was to evaluate the effectiveness of initiating opiate replacement therapy prior to release from incarceration on reducing HIV risk behaviors and drug relapse. In addition, this study evaluated the effectiveness of short-term payment versus non-payment of community opiate replacement therapy immediately following release from incarceration.

DETAILED DESCRIPTION:
A substantial proportion of individuals addicted to heroin are incarcerated while addicted and a majority of individuals released from a correctional setting have a history of heroin addiction. The period immediately after release from incarceration is a particularly high-risk time for HIV transmission and other problems, including drug relapse and overdose. Methadone treatment is the most widely used opiate replacement therapy in the United States and has been shown to decrease HIV risk, as well as drug use, addiction relapse, and criminal activity. The purpose of this study was to evaluate the effectiveness of initiating opiate replacement therapy prior to release from incarceration on reducing HIV risk behaviors and drug relapse. In addition, this study evaluated the effectiveness of short-term payment versus non-payment of community opiate replacement therapy immediately following release from incarceration.

Participants in this were randomly assigned to 1 of 3 treatment groups. Participants enrolled in Group 1 initiated methadone opiate replacement therapy about 1 month prior to release from incarceration. They proceeded with a methadone program of their choice upon release and received short-term payment to cover treatment costs. Participants enrolled in Group 2 were referred to a methadone program of their choice and received short-term payment to cover treatment costs. Participants enrolled in Group 3 were referred to a program of choice upon release from incarceration without receiving financial assistance. All participants had the opportunity to partake in existing support programs available at the Rhode Island Department of Corrections while incarcerated and in the community upon release. Follow-up assessments occurred at Months 1.5, 6, and 12. These included interviews and urine specimens for toxicology analysis to verify self-reports.

ELIGIBILITY:
Inclusion Criteria:

* Currently incarcerated at the Rhode Island Department of Corrections with a scheduled release date at least 28 days after enrollment
* Incarceration length not to have exceeded two years at the time of enrollment
* Heroin dependent with self-reported heroin injection in the month prior to incarceration OR enrollment in a methadone treatment program prior to incarceration for heroin addiction with a history of injection drug use
* Desire to enter methadone treatment upon release and plans to secure funding for methadone treatment after study completion
* History of prior tolerance to methadone
* History of at least one drug-related incarceration
* Speaks English or Spanish
* Plans to remain in Rhode Island for the duration of the study (24 months)
* Ability to provide at least two names of individuals who can verify participant information

Exclusion Criteria:

* Currently receiving methadone at the Rhode Island Department of Corrections
* Currently undergoing a non-narcotic detoxification from illicit opiates at the Rhode Island Department of Corrections
* Plans to leave Rhode Island within the two years following enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josiah D Rich, M.P.H., M.D., Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment occurred at the Rhode Island Department of Corrections. Screening began on 9/15/2006 and the first participant was enrolled on 9/29/2006. The last participant was enrolled on 2/20/2009.
Pre-assignment Details: There were no significant events following participant enrollment and prior to group assignment.
Groups:
- Pre-release MMT Initiation + Referral Post Release + Payment: Participants assigned to this arm will undergo extensive assessment (physical, medical history, drug use and treatment history) prior to initiating treatment. MMT will begin 1-30 days prior to release from incarceration. MMT first dose will begin at 5 mg with 2 mg increase per day until release or therapeutic dose of 60-120 mg is achieved. Daily observation by dosing nurses and twice weekly symptom review by Research Assistant will occur. Additionally, participants assigned to Arm 1 will have all logistical arrangements made for entry into a community methadone clinic program within 24 hours of release from incarceration. The study will fully pay for MMT for 12 weeks and half the costs of treatment for the next 12 weeks.
- MMT Referral Post Release + Payment: Participants assigned to this arm will have all logistical arrangements made for entry into a community methadone clinic program within 24-48 hours of release from incarceration. The study will fully pay for MMT for 12 weeks and half the costs of treatment for the next 12 weeks.
- MMT Referral Post Release: Participants assigned to this arm will not begin treatment prior to release from incarceration or have treatment paid for by the study. However, study staff will work with participants to identify ways to pay for treatment, including assisting with Medicaid applications, etc. Further, the study will make the logistical arrangements for entering treatment if participant has a means to finance MMT.
Period: Overall Study
Arm/Group | Pre-release MMT Initiation + Referral Post Release + Payment | MMT Referral Post Release + Payment | MMT Referral Post Release
Started | 29 | 28 | 30
Completed | 26 | 20 | 23
Not Completed | 3 | 8 | 7
Not completed — Other reason | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 5 | 5
Not completed — Death | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pre-release MMT Initiation + Referral Post Release + Payment: Participants enrolled in Group 1 will initiate methadone opiate replacement therapy about 1 month prior to release from incarceration. They will then proceed with a methadone program of choice upon release and receive short-term payment to cover treatment costs.
- MMT Referral Post Release + Payment: Participants enrolled in Group 2 will be referred to a methadone program of choice upon release from incarceration with provision of short-term payment of treatment costs.
- MMT Referral Post Release: Participants enrolled in Group 3 will be referred to a program of their choice upon release from incarceration without receiving financial assistance.
- Total: Total of all reporting groups
Arm/Group | Pre-release MMT Initiation + Referral Post Release + Payment | MMT Referral Post Release + Payment | MMT Referral Post Release | Total
Number analyzed (Participants) | 29 | 28 | 30 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 28 | 30 | 87
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (8.79) | 37 (6.69) | 38.4 (9.25) | 37.6 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 9 | 27
  Male | 19 | 20 | 21 | 60
Region of Enrollment [Number; unit: participants]
  United States | 29 | 28 | 30 | 87

OUTCOME MEASURES:

1. Primary Outcome: Treatment Engagement
Description: Participants are considered to have successfully initiated community methadone maintenance treatment only if they make their first clinic appointment within 30 days after being released from incarceration. This outcome is measured by frequency - yes, participant attended initial clinic appointment within 30 days post release or no, participant did not attend clinic appointment within 30 days post release. Data source was methadone clinic chart review.
Time Frame: within 30 days post release of incarceration
Population: We assessed community methadone treatment clinic attendance of all enrolled participants based on clinic chart review.
Measure: Number; unit: participants
Groups:
- As Assigned: Pre-release MMT + Referral Post Release + Payment: Participants enrolled in Group 1 will initiate methadone opiate replacement therapy about 1 month prior to release from incarceration. They will be linked to a methadone treatment program of their choice upon release from incarceration with provision of short-term payment of treatment costs.
- As Assigned: MMT Referral Post Release + Payment: Participants enrolled in Group 2 will be linked to a methadone treatment program of their choice upon release from incarceration with provision of short-term payment of treatment costs.
- As Assigned: MMT Referral Post Release: Participants enrolled in Group 3 will be referred to a methadone program of their choice upon release from incarceration without receiving financial assistance.
Arm/Group | As Assigned: Pre-release MMT + Referral Post Release + Payment | As Assigned: MMT Referral Post Release + Payment | As Assigned: MMT Referral Post Release
Number analyzed (Participants) | 29 | 28 | 30
participants | 23 | 11 | 6
Statistical Analysis 1: Comparison: As Assigned: Pre-release MMT + Referral Post Release + Payment vs As Assigned: MMT Referral Post Release + Payment vs As Assigned: MMT Referral Post Release; Outcome: engage in treatment post release, yes or no; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected

2. Primary Outcome: Time to MMT Initiation Post Release Based on Clinic Chart Review
Description: Participants are considered to have successfully initiated community methadone maintenance treatment only if they make their first clinic appointment within 30 days after being released from incarceration. This outcome measures number of days from release to the first day of clinic attendance, only for those participants who successfully entered methadone treatment post release. Data source was methadone clinic chart review.
Time Frame: within 30 days post release from incarceration
Population: Participants were analyzed as randomized (intent to treat). We calculated the mean number of days (and SD) between release from incarceration and first MMT clinic visit post release. Not all participants attended clinic within 30 days post release - those participants are not included in this analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | As Assigned: Pre-release MMT + Referral Post Release + Payment | As Assigned: MMT Referral Post Release + Payment | As Assigned: MMT Referral Post Release
Number analyzed (Participants) | 23 | 11 | 6
days | 2 (4.37) | 9 (9.74) | 5 (5.16)
Statistical Analysis 1: Comparison: As Assigned: Pre-release MMT + Referral Post Release + Payment vs As Assigned: MMT Referral Post Release + Payment vs As Assigned: MMT Referral Post Release; Test type: Superiority or Other; p = .02, Chi-squared, Corrected

3. Primary Outcome: HIV Risk Behaviors - Self Report
Description: Participants who self-reported injecting illicit drugs in the past 30 days, based on responses to face-to-face administration of the 6 month interview.
Time Frame: 6 month follow-up interviews
Measure: Number; unit: participants
Groups:
- As Assigned: Pre-release MMT + Referral Post Release + Payment: Participants enrolled in Group 1 will initiate methadone opiate replacement therapy about 1 month prior to release from incarceration. They will then proceed with a methadone program of choice upon release and receive short-term payment to cover treatment costs.
- As Assigned: MMT Referral Post Release + Payment: Participants enrolled in Group 2 will be referred to a methadone program of choice upon release from incarceration with provision of short-term payment of treatment costs.
- As Assigned: MMT Referral Post Release: Participants enrolled in Group 3 will be referred to a program of their choice upon release from incarceration without receiving financial assistance.
Arm/Group | As Assigned: Pre-release MMT + Referral Post Release + Payment | As Assigned: MMT Referral Post Release + Payment | As Assigned: MMT Referral Post Release
Number analyzed (Participants) | 25 | 16 | 21
participants | 3 | 6 | 8
Statistical Analysis 1: Comparison: As Assigned: Pre-release MMT + Referral Post Release + Payment vs As Assigned: MMT Referral Post Release + Payment vs As Assigned: MMT Referral Post Release; Test type: Superiority or Other; p = .09, Chi-squared, Corrected

4. Secondary Outcome: Drug Use
Description: Participants who self-reported heroin use in the past 30 days, based on responses to face-to-face administration of the 6 month interview.
Time Frame: 6 month follow-up interviews
Measure: Number; unit: participants
Groups:
- As Assigned: MMT Pre-release + Referral Post Release + Payment: Participants enrolled in Group 1 will initiate methadone opiate replacement therapy about 1 month prior to release from incarceration. They will then proceed with a methadone program of choice upon release and receive short-term payment to cover treatment costs.
Arm/Group | As Assigned: MMT Pre-release + Referral Post Release + Payment | As Assigned: MMT Referral Post Release + Payment | As Assigned: MMT Referral Post Release
Number analyzed (Participants) | 25 | 16 | 21
participants | 6 | 8 | 11
Statistical Analysis 1: Comparison: As Assigned: MMT Pre-release + Referral Post Release + Payment vs As Assigned: MMT Referral Post Release + Payment vs As Assigned: MMT Referral Post Release; Test type: Superiority or Other; p = .09, Chi-squared, Corrected

5. Secondary Outcome: Fatal Overdose
Description: Number of participants who died as the result of drug poisoning within six months of release of incarceration. This outcome was based on review of death records.
Time Frame: Within six months from release of incarceration
Measure: Number; unit: participants
Arm/Group | As Assigned: MMT Pre-release + Referral Post Release + Payment | As Assigned: MMT Referral Post Release + Payment | As Assigned: MMT Referral Post Release
Number analyzed (Participants) | 29 | 28 | 30
participants | 0 | 1 | 1

6. Secondary Outcome: Non-fatal Overdose
Description: Participants who self-reported experiencing an overdose within the past six months, based on responses to face-to-face administration of the 6 month interview.
Time Frame: 6 month follow-up interviews
Measure: Number; unit: participants
Arm/Group | As Assigned: MMT Pre-release + Referral Post Release + Payment | As Assigned: MMT Referral Post Release + Payment | As Assigned: MMT Referral Post Release
Number analyzed (Participants) | 25 | 16 | 21
participants | 3 | 3 | 2
Statistical Analysis 1: Comparison: As Assigned: MMT Pre-release + Referral Post Release + Payment vs As Assigned: MMT Referral Post Release + Payment vs As Assigned: MMT Referral Post Release; Test type: Superiority or Other; p = 0.8, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: 12 months
Description: Fatal Overdoses
Groups:
- As Assigned: Pre-release MMT + Referral Post Release + Payment: Participants enrolled in Group 1 will initiate methadone opiate replacement therapy about 1 month prior to release from incarceration. They will then proceed with a methadone program of choice upon release and receive short-term payment to cover treatment costs.
  Fatal overdose deaths are calculated using all participants assigned to Arm 1. Other adverse events are calculated using self reported data from 12 month interviews.
- As Assigned: MMT Referral Post Release + Payment: Participants enrolled in Group 2 will be referred to a methadone program of choice upon release from incarceration with provision of short-term payment of treatment costs.
  Fatal overdose deaths are calculated using all participants assigned to Arm 2. Other adverse events are calculated using self reported data from 12 month interviews.
- As Assigned: MMT Referral Post Release: Participants enrolled in Group 3 will be referred to a program of their choice upon release from incarceration without receiving financial assistance.
  Fatal overdose deaths are calculated using all participants assigned to Arm 3. Other adverse events are calculated using self reported data from 12 month interviews.
Arm/Group | As Assigned: Pre-release MMT + Referral Post Release + Payment | As Assigned: MMT Referral Post Release + Payment | As Assigned: MMT Referral Post Release
Serious Adverse Events (participants affected / at risk) | 0/29 | 2/28 | 1/30
Other Adverse Events (participants affected / at risk) | 10/26 | 8/20 | 8/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | As Assigned: Pre-release MMT + Referral Post Release + Payment (N=29) | As Assigned: MMT Referral Post Release + Payment (N=28) | As Assigned: MMT Referral Post Release (N=30)
Fatal Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | As Assigned: Pre-release MMT + Referral Post Release + Payment (N=26) | As Assigned: MMT Referral Post Release + Payment (N=20) | As Assigned: MMT Referral Post Release (N=23)
Non-fatal Overdose (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 2 (2) — Any overdose reported by participants in the 12 month post release interview. These were not related to participation in the study.
ER visits (Injury, poisoning and procedural complications) | 10 (10) | 7 (7) | 7 (7) — Any ER visits that were reported by participants in the 12 month post release interview. These were not related to participation in the study.
Hospitalizations (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1) — Any hospitalizations that were reported by participants in the 12 month post release interview. These were not related to participation in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No